CLINICAL TRIAL: NCT03582631
Title: Biomarkers in Acute High-risk AbdoMinAl Surgery
Acronym: BAHAMAS
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Rune Børch Hasselager, Principal Investigator, Medical Doctor, University of Copenhagen
Other Study IDs: BAHAMAS1
Record Dates: First submitted 2018-06-11; First posted 2018-07-11 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: General Surgery; Inflammation; Troponins; Biomarkers
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples were collected at the time of induction of anaesthesia. For AHA-patients a pre-operative optimisation protocol was introduced in the hospital throughout the data collection period, which stated that the patient was optimized with goal directed fluid therapy before induction of anaesthesia. The blood samples were usually taken from the arterial line used for invasive blood pressure monitoring but some were obtained from venous puncture with standard preoperative tests.
  The blood samples were collected in tubes with EDTA as anti-coagulant for plasma and in tubes with coagulation enhancer for serum. After centrifugation for 10 mins at room temperature the plasma and serum, respectively were transferred to freezing tubes for subsequent long-term storage at -80C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Emergency abdominal surgery — Emergency surgery for high-risk abdominal pathology using a protocol for optimized perioperative care

SUMMARY:
Acute high-risk abdominal surgery (AHA) is performed in hospitals worldwide. Ethiologies are heterogeneous, but it carries a high mortality rate (1)(2). In particular, emergency laparotomies performed on elderly people has a high mortality rate(3)(4). Different quality improvement programs have been suggested, but the quality of care and mortality varies between hospitals (5)(6). The use of postoperative intensive care seem to be inadequate for this high risk population (1)(7)(8). It is of paramount importance to identify the frailest and acutely deranged patients, who are in risk of poor outcome, to allocate resources for optimization postoperatively. Failure to escalate care intensity after having developed postoperative complications affect outcome. Organization, teamwork and culture is important postoperatively to be able to escalate care especially in standard care wards (9)(10). However, it is difficult to predict which patients will develop complications.

Different risk assessment tools have been proposed for patients undergoing AHA (11)(12). The APACHE-II score, even though developed for critical care, seems to give the best prediction of outcome. Objective risk assessment tools support clinical decision making as subjective clinical assessment often underestimates the risk for the patients in highest risk of complications and death (13). Good clinical decision-making is likely to improve the clinical outcome by allocating appropriate resources. Prognostic tools are also useful to inform patients about what to expect in the postoperative phase and of long-term outcome. Especially in the elder population with increased risk of loss of function or independency, this can be useful to give informed consent to treatment. Furthermore, good risk assessment is important to optimize palliative care after end-of-life decisions, which is often ignored in research, but highly relevant in clinical work.

Prognostic biomarkers in other high mortality populations have received much attention for risk stratification (14). An ideal biomarker should be readily available upon decision-making, easy to measure, and reliable. Furthermore, it should accurately differentiate prognosis for patients to have value in the clinical decision-making and guide the treatment. It should also be linked to the clinical outcomes.

The investigators aim to identify AHA biomarkers that are prognostic or predictive for postoperative morbidity, mortality and length of hospitalization.

DETAILED DESCRIPTION:
Acute high-risk abdominal surgery (AHA) is performed in hospitals worldwide. Ethiologies are heterogeneous, but overall emergency surgery carries a very high mortality rate (1)(2). In particular, emergency laparotomies performed on elderly people has a high mortality rate(3)(4). Different quality improvement programmes for that particular patient group have been suggested, but the quality of care and thereby mortality varies considerably between hospitals(5)(6). The use of postoperative intensive care and monitoring seem to be inadequate for this high risk population in a variety of hospitals(1)(7)(8). It is of paramount importance to identify the frailest and most acutely deranged patients, who are in risk of poor outcome, in order to allocate resources for improved monitoring and optimisation postoperatively. It has been shown that failure to rescue patients after having developed postoperative complications and inability to escalate care intensity affects the outcome. Organisation, teamwork and culture is important in the postoperative phase to be able to escalate care especially in standard care wards(9)(10). However, it is found difficult to predict which patients will experience complications in a standard care ward.

Different risk assessment tools have been proposed for patients undergoing AHA(11)(12). The APACHE-II score, even though developed for critical care, seems to be the one with best prediction of outcome. Risk assessment tools are important to support clinical decision making by the perioperative team as subjective clinical assessment often underestimates the risk for the patients in highest risk of complications and death(13). Good clinical decision-making is likely to improve the clinical outcome by allocating appropriate resources. Prognostic tools are also useful to inform patients about what to expect in the immediate postoperative phase and of long-term outcome. Especially in the elder population with increased risk of long hospitalisation and loss of function or independency this can be useful to give informed consent to treatment strategy. Furthermore, good risk assessment is important to optimize palliative care after end-of-life decisions, which is often ignored in research, but highly relevant in clinical work.

During recent years use of prognostic biomarkers in other high mortality populations have received much attention for risk stratification(14). An ideal biomarker should be readily available upon decision-making, easy to measure, reliable and biologically stable. Furthermore it has to be able to accurately differentiate prognosis for patients to have value in the clinical decision-making and guide the treatment of the patient. It should be linked to the clinical outcomes.

The investigators aim to identify serological AHA biomarkers that are prognostic or predictive for postoperative morbidity, mortality and length of hospitalisation.

Data collection Data on mortality was obtained using the Danish Civil Registration System(30). This register is maintained by the Danish government and assigns a unique personal identification number to all Danish citizens. It contains data on address, immigration emigration, gender, date of birth and exact day of death. It is updated within days of any change in information.

Other data were collected in the medical records of patients. Complications were defined using the Clavien-Dindo Classification for Surgical Complications(31).

Outcome measures Primary outcomes are short and long-term mortality (30 days and 180 days respectively) and major complications during index hospitalization (Clavien-Dindo >2). Secondary outcomes are length of hospitalisation, length of intensive care admission as well as perioperative need for inotropic or vasopressor support and high volume fluid resuscitation.

Description of biological material Blood samples were collected at the time of induction of anaesthesia. For AHA-patients a pre-operative optimisation protocol was introduced in the hospital throughout the data collection period, which stated that the patient was optimized with goal directed fluid therapy before induction of anaesthesia. The blood samples were usually taken from the arterial line used for invasive blood pressure monitoring but some were obtained from venous puncture with standard preoperative tests.

The blood samples were collected in tubes with EDTA as anti-coagulant for plasma and in tubes with coagulation enhancer for serum. After centrifugation for 10 mins at room temperature the plasma and serum, respectively were transferred to freezing tubes for subsequent long-term storage at -80C.

Limitations of the study Data collection during clinical work including blood samples requires resources and is susceptible to selection and information bias. It is possible that resources for collecting blood samples correctly where reduced for the most unstable patients at the time of induction of anaesthesia. Patients who were considered too frail to undergo surgery, where a palliative or conservative approach was chosen, were not included in this study. Postoperatively, patients in the AHA-cohort were assigned to postoperative intensive monitoring in the post-operative care unit if they had American Society of Anaesthesiologist physical performance score(34) above two. This stratification is susceptible to information-bias because of inter-observer variation(35).

The data is collected in a single medical facility with and optimized care protocol for AHA and can therefore not uncritically be applied to other populations.

Economical support and budget:

The clinical study as well as establishment of the biobank has been supported by a grant from the Capital Region of Denmark (Region H). The cost of biochemical analysis will be covered by the Department of Clinical Biochemistry, Hvidovre Hospital. Other expenses will be covered by the AHA research group, Department of Anaesthesiology and Intensive Care and Department of Surgical Gastroenterology, Hvidovre Hospital.

Publication of results:

Results from the studies will be published in medical journals indexed in the PubMed/EMBASE database.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older with the suspicion for abdominal pathology requiring immediate emergency laparotomy or laparoscopy including reoperations after elective surgery and reoperations after previous AHA surgery.

Exclusion Criteria:

* We excluded the following procedures: appendectomies; negative laparoscopies and laparotomies; cholecystectomies; simple herniotomies following incarceration (without intestinal resection); reoperation due to fascial separation with no other abdominal pathology; internal herniation after roux-en-y gastric bypass surgery; sub-acute surgery (planned within 48 hours) for inflammatory bowel disease; and sub-acute colorectal cancer surgery.

We excluded, traumas, pregnant woman, uro-genital, gynaecological and vascular pathology except for mesenteric ischemia.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Include patients with a preoperative blood sample stored in the bio bank; the patients did undergo AHA at Hvidovre Hospital, Copenhagen, Denmark, from June 1st 2013 when the AHA study protocol was initiated.
  In the primary study we will include the first 100 consecutive primary operations in the cohort.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
No of patients died within 30 days postoperatively | 30 days
  30 day mortality after surgery
No of patients died within 180 days postoperatively | 180 days
  180-day mortality after surgery
No of patients with major postoperative complications within 30 days afer surgery | 30 days
  Clavien Dindo grade more than 3a

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai B Foss, DMSc, Principal Investigator — Department of Anaesthesiology, Hvidovre University Hospital, Denmark
Locations (1):
- Hvidovre University hospital, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Tolstrup MB, Watt SK, Gogenur I. Morbidity and mortality rates after emergency abdominal surgery: an analysis of 4346 patients scheduled for emergency laparotomy or laparoscopy. Langenbecks Arch Surg. 2017 Jun;402(4):615-623. doi: 10.1007/s00423-016-1493-1. Epub 2016 Aug 9. PMID 27502400
- [Background] Stoneham M, Murray D, Foss N. Emergency surgery: the big three--abdominal aortic aneurysm, laparotomy and hip fracture. Anaesthesia. 2014 Jan;69 Suppl 1:70-80. doi: 10.1111/anae.12492. PMID 24303863
- [Background] Jeppesen MH, Tolstrup MB, Kehlet Watt S, Gogenur I. Risk factors affecting morbidity and mortality following emergency laparotomy for small bowel obstruction: A retrospective cohort study. Int J Surg. 2016 Apr;28:63-8. doi: 10.1016/j.ijsu.2016.02.059. Epub 2016 Feb 18. PMID 26912017
- [Background] Saunders DI, Murray D, Pichel AC, Varley S, Peden CJ; UK Emergency Laparotomy Network. Variations in mortality after emergency laparotomy: the first report of the UK Emergency Laparotomy Network. Br J Anaesth. 2012 Sep;109(3):368-75. doi: 10.1093/bja/aes165. Epub 2012 Jun 22. PMID 22728205
- [Background] Symons NR, Moorthy K, Almoudaris AM, Bottle A, Aylin P, Vincent CA, Faiz OD. Mortality in high-risk emergency general surgical admissions. Br J Surg. 2013 Sep;100(10):1318-25. doi: 10.1002/bjs.9208. Epub 2013 Jul 17. PMID 23864490
- [Background] Jhanji S, Thomas B, Ely A, Watson D, Hinds CJ, Pearse RM. Mortality and utilisation of critical care resources amongst high-risk surgical patients in a large NHS trust. Anaesthesia. 2008 Jul;63(7):695-700. doi: 10.1111/j.1365-2044.2008.05560.x. Epub 2008 May 16. PMID 18489613
- [Background] Vester-Andersen M, Lundstrom LH, Moller MH, Waldau T, Rosenberg J, Moller AM; Danish Anaesthesia Database. Mortality and postoperative care pathways after emergency gastrointestinal surgery in 2904 patients: a population-based cohort study. Br J Anaesth. 2014 May;112(5):860-70. doi: 10.1093/bja/aet487. Epub 2014 Feb 10. PMID 24520008
- [Background] Johnston MJ, Arora S, King D, Bouras G, Almoudaris AM, Davis R, Darzi A. A systematic review to identify the factors that affect failure to rescue and escalation of care in surgery. Surgery. 2015 Apr;157(4):752-63. doi: 10.1016/j.surg.2014.10.017. PMID 25794627
- [Background] Ghaferi AA, Dimick JB. Importance of teamwork, communication and culture on failure-to-rescue in the elderly. Br J Surg. 2016 Jan;103(2):e47-51. doi: 10.1002/bjs.10031. Epub 2015 Nov 30. PMID 26616276
- [Background] Oliver CM, Walker E, Giannaris S, Grocott MP, Moonesinghe SR. Risk assessment tools validated for patients undergoing emergency laparotomy: a systematic review. Br J Anaesth. 2015 Dec;115(6):849-60. doi: 10.1093/bja/aev350. Epub 2015 Nov 3. PMID 26537629
- [Background] Al-Temimi MH, Griffee M, Enniss TM, Preston R, Vargo D, Overton S, Kimball E, Barton R, Nirula R. When is death inevitable after emergency laparotomy? Analysis of the American College of Surgeons National Surgical Quality Improvement Program database. J Am Coll Surg. 2012 Oct;215(4):503-11. doi: 10.1016/j.jamcollsurg.2012.06.004. Epub 2012 Jul 11. PMID 22789546
- [Background] Hobson SA, Sutton CD, Garcea G, Thomas WM. Prospective comparison of POSSUM and P-POSSUM with clinical assessment of mortality following emergency surgery. Acta Anaesthesiol Scand. 2007 Jan;51(1):94-100. doi: 10.1111/j.1399-6576.2006.01167.x. Epub 2006 Nov 1. PMID 17073858
- [Background] Sandquist M, Wong HR. Biomarkers of sepsis and their potential value in diagnosis, prognosis and treatment. Expert Rev Clin Immunol. 2014 Oct;10(10):1349-56. doi: 10.1586/1744666X.2014.949675. Epub 2014 Aug 21. PMID 25142036
- [Background] Donadello K, Scolletta S, Taccone FS, Covajes C, Santonocito C, Cortes DO, Grazulyte D, Gottin L, Vincent JL. Soluble urokinase-type plasminogen activator receptor as a prognostic biomarker in critically ill patients. J Crit Care. 2014 Feb;29(1):144-9. doi: 10.1016/j.jcrc.2013.08.005. Epub 2013 Oct 9. PMID 24120089
- [Background] Liu X, Shen Y, Li Z, Fei A, Wang H, Ge Q, Pan S. Prognostic significance of APACHE II score and plasma suPAR in Chinese patients with sepsis: a prospective observational study. BMC Anesthesiol. 2016 Jul 29;16(1):46. doi: 10.1186/s12871-016-0212-3. PMID 27473112
- [Background] Zeng M, Chang M, Zheng H, Li B, Chen Y, He W, Huang C. Clinical value of soluble urokinase-type plasminogen activator receptor in the diagnosis, prognosis, and therapeutic guidance of sepsis. Am J Emerg Med. 2016 Mar;34(3):375-80. doi: 10.1016/j.ajem.2015.11.004. Epub 2015 Nov 9. PMID 26615223
- [Background] Donadello K, Scolletta S, Covajes C, Vincent JL. suPAR as a prognostic biomarker in sepsis. BMC Med. 2012 Jan 5;10:2. doi: 10.1186/1741-7015-10-2. PMID 22221662
- [Background] Hodges GW, Bang CN, Wachtell K, Eugen-Olsen J, Jeppesen JL. suPAR: A New Biomarker for Cardiovascular Disease? Can J Cardiol. 2015 Oct;31(10):1293-302. doi: 10.1016/j.cjca.2015.03.023. Epub 2015 Mar 25. PMID 26118447
- [Background] Botha S, Fourie CMT, Schutte R, Eugen-Olsen J, Pretorius R, Schutte AE. Soluble urokinase plasminogen activator receptor as a prognostic marker of all-cause and cardiovascular mortality in a black population. Int J Cardiol. 2015 Apr 1;184:631-636. doi: 10.1016/j.ijcard.2015.03.041. Epub 2015 Mar 4. PMID 25771228
- [Background] Sando A, Schultz M, Eugen-Olsen J, Rasmussen LS, Kober L, Kjoller E, Jensen BN, Ravn L, Lange T, Iversen K. Introduction of a prognostic biomarker to strengthen risk stratification of acutely admitted patients: rationale and design of the TRIAGE III cluster randomized interventional trial. Scand J Trauma Resusc Emerg Med. 2016 Aug 5;24:100. doi: 10.1186/s13049-016-0290-8. PMID 27491822
- [Background] Lahiri R, Derwa Y, Bashir Z, Giles E, Torrance HD, Owen HC, O'Dwyer MJ, O'Brien A, Stagg AJ, Bhattacharya S, Foster GR, Alazawi W. Systemic Inflammatory Response Syndrome After Major Abdominal Surgery Predicted by Early Upregulation of TLR4 and TLR5. Ann Surg. 2016 May;263(5):1028-37. doi: 10.1097/SLA.0000000000001248. PMID 26020106
- [Background] John J, Woodward DB, Wang Y, Yan SB, Fisher D, Kinasewitz GT, Heiselman D. Troponin-I as a prognosticator of mortality in severe sepsis patients. J Crit Care. 2010 Jun;25(2):270-5. doi: 10.1016/j.jcrc.2009.12.001. Epub 2010 Feb 10. PMID 20149590
- [Background] Landesberg G, Jaffe AS, Gilon D, Levin PD, Goodman S, Abu-Baih A, Beeri R, Weissman C, Sprung CL, Landesberg A. Troponin elevation in severe sepsis and septic shock: the role of left ventricular diastolic dysfunction and right ventricular dilatation*. Crit Care Med. 2014 Apr;42(4):790-800. doi: 10.1097/CCM.0000000000000107. PMID 24365861
- [Background] Sheyin O, Davies O, Duan W, Perez X. The prognostic significance of troponin elevation in patients with sepsis: a meta-analysis. Heart Lung. 2015 Jan-Feb;44(1):75-81. doi: 10.1016/j.hrtlng.2014.10.002. Epub 2014 Nov 18. PMID 25453390
- [Background] Benz F, Roy S, Trautwein C, Roderburg C, Luedde T. Circulating MicroRNAs as Biomarkers for Sepsis. Int J Mol Sci. 2016 Jan 9;17(1):78. doi: 10.3390/ijms17010078. PMID 26761003
- [Background] Johansson PI, Stensballe J, Rasmussen LS, Ostrowski SR. A high admission syndecan-1 level, a marker of endothelial glycocalyx degradation, is associated with inflammation, protein C depletion, fibrinolysis, and increased mortality in trauma patients. Ann Surg. 2011 Aug;254(2):194-200. doi: 10.1097/SLA.0b013e318226113d. PMID 21772125
- [Background] Nemeth E, Rivera S, Gabayan V, Keller C, Taudorf S, Pedersen BK, Ganz T. IL-6 mediates hypoferremia of inflammation by inducing the synthesis of the iron regulatory hormone hepcidin. J Clin Invest. 2004 May;113(9):1271-6. doi: 10.1172/JCI20945. PMID 15124018
- [Background] Gallo V, Egger M, McCormack V, Farmer PB, Ioannidis JP, Kirsch-Volders M, Matullo G, Phillips DH, Schoket B, Stromberg U, Vermeulen R, Wild C, Porta M, Vineis P; STROBE Statement. STrengthening the Reporting of OBservational studies in Epidemiology--Molecular Epidemiology (STROBE-ME): an extension of the STROBE Statement. PLoS Med. 2011 Oct;8(10):e1001117. doi: 10.1371/journal.pmed.1001117. Epub 2011 Oct 25. PMID 22039356
- [Background] Pedersen CB. The Danish Civil Registration System. Scand J Public Health. 2011 Jul;39(7 Suppl):22-5. doi: 10.1177/1403494810387965. PMID 21775345
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Sankar A, Johnson SR, Beattie WS, Tait G, Wijeysundera DN. Reliability of the American Society of Anesthesiologists physical status scale in clinical practice. Br J Anaesth. 2014 Sep;113(3):424-32. doi: 10.1093/bja/aeu100. Epub 2014 Apr 11. PMID 24727705

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT03582631/Prot_SAP_001.pdf